CLINICAL TRIAL: NCT01958593
Title: A Randomized, Double-Blind, Controlled Phase 2 Pilot Study of Manualized 3,4-methylenedioxymethamphetamine (MDMA)-Assisted Psychotherapy in 12 Subjects With Treatment-Resistant Posttraumatic Stress Disorder (PTSD) - Canada
Brief Title: Randomized, Double-blind, Controlled of MDMA-assisted Psychotherapy in 12 Subjects With PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This pilot study was terminated early by sponsor due to insufficient rate of accrual.
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MP-4
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic stress disorder; MDMA; psychotherapy; therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo with therapy (Placebo Comparator): Participants will receive placebo with therapy during each of two experimental sessions.
  Interventions: Drug: Placebo; Behavioral: Psychotherapy
- MDMA-assisted therapy (Experimental): Participants will receive MDMA (initial dose of 125 mg midomafetamine HCl followed by a supplemental dose of 62.5 mg midomafetamine HCl) with therapy during each of two experimental sessions.
  Interventions: Drug: Midomafetamine HCl; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Placebo — Placebo with therapy administered in two blinded experimental sessions. Participants in this group in Stage 1 may take part in Stage 2.
  Other Names: Inactive placebo
  Arms: Placebo with therapy
Drug: Midomafetamine HCl — Participants will receive MDMA-assisted therapy during two blinded experimental sessions. After unblinding, may receive a third session of open-label MDMA-assisted therapy.
  Other Names: MDMA HCl; 3,4-methylenedioxymethamphetamine; midomafetamine; MDMA
  Arms: MDMA-assisted therapy
Behavioral: Psychotherapy — Psychotherapy before and after experimental sessions.

SUMMARY:
The goal of this clinical trial is to compare full dose MDMA-assisted therapy to placebo with therapy in participants with chronic, treatment-resistant PTSD. The main question it aims to answer is: Does MDMA-assisted therapy versus placebo with therapy reduce PTSD symptoms?

Participants will receive either MDMA-assisted therapy or placebo with therapy during two blinded experimental sessions spaced three to five weeks apart. During experimental sessions, participants receive an initial dose of 125 mg of MDMA HCl, or placebo, followed by a dose of 62.5 mg of MDMA HCl, or placebo. During this treatment period, participants will also undergo non-drug preparatory therapy sessions and non-drug integration sessions.

Researchers will compare PTSD symptoms in the MDMA-assisted therapy group to the placebo with therapy group to see if there is a reduction in symptoms after the treatment period. Safety measures will also be assessed between groups.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical study will assess the safety and efficacy of MDMA-assisted therapy in treating chronic, treatment-resistant PTSD. In Stage 1, participants will be randomized to either MDMA-assisted therapy or placebo with therapy during two blinded experimental sessions, spaced three to five weeks apart. During experimental sessions, participants receive an initial dose of 125 mg of MDMA HCl, or placebo, followed by a dose of 62.5 mg of MDMA HCl, or placebo. During this treatment period, participants will also undergo non-drug preparatory therapy sessions and non-drug integration sessions. After this treatment period, participants will complete the primary endpoint assessment and the study will become unblinded.

Participants who were assigned to receive MDMA-assisted therapy will receive a third session of MDMA-assisted therapy that is open-label and participants assigned to receive placebo with therapy will have the option to enter Stage 2. Stage 2 will explore the optimal therapeutic dose of MDMA in a clinical titration dosing strategy. Participants will receive MDMA-assisted with an initial dose of 100 mg followed by a dose of 50 mg of MDMA HCl for the first experimental session. In the second and third experimental sessions, participants will have the option to increase the dose to an initial dose of 125 mg followed by a dose of 62.5 mg.

A blinded independent rater will assess PTSD symptoms via the CAPS-IV as well as other secondary outcome measures and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe PTSD;
* Have chronic PTSD, defined as persisting for longer than 6 months;
* Have treatment-resistant PTSD, meaning unable to achieve remission despite previous therapy or medication or discontinued treatment due to inability to tolerate previous therapy or medication;
* Are willing to refrain from taking any psychiatric medications during the study period;
* Willing to remain overnight at the study site;
* Agree to have transportation home after experimental sessions;
* Are willing to be contacted via telephone for all necessary telephone contacts;
* Must have a negative pregnancy test if able to bear children, and agree to use an effective form of birth control;
* Are proficient in speaking and reading English;
* Agree not to participate in any other interventional clinical trials during the duration of this study.

Exclusion Criteria:

* Are pregnant or nursing, or if of child bearing potential, are not practicing an effective means of birth control;
* Weigh less than 48 kg;
* Are unable to give adequate informed consent;
* Upon review of past and current drugs/medication must not be on or have taken a medication that is exclusionary;
* Have used "Ecstasy" (illicit drug preparations purported to contain MDMA) more than five times in the last 10 years or at least once within six months of enrollment;
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Pacey, MBBS FRCP[C], Principal Investigator — University of Victoria
Locations (1):
- Offices of Dr. Ingrid Pacey MBBS FRCP[C], Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through printed ads, internet ads, referrals from other psychiatrists, psychotherapists or physicians, and through word of mouth.
Groups:
- MDMA-assisted Therapy: Participants will receive full-dose (125 mg) MDMA with therapy during each of two experimental sessions.
Period: Stage 1
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Started | 2 | 4
Completed (Primary Endpoint) | 2 | 4
Not Completed | 0 | 0
Period: Stage 2 Open-label Crossover
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Started (Stage 2 open-label crossover included only those participants assigned placebo in Stage 1) | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo With Therapy: Participants will receive placebo with therapy during each of two blinded experimental sessions.
- MDMA-assisted Therapy: Participants will receive MDMA-assisted therapy during each of two blinded experimental sessions.
- Total: Total of all reporting groups
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.66) | 49.6 (7.9) | 47.7 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2 | 3 | 5
  Race: Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS-IV) Score From Baseline to Primary Endpoint
Description: Clinician-administered and scored assessment of PTSD symptoms via structured interview, including global symptom severity, dichotomous diagnostic score and subscale scores. The Clinician-Administered PTSD Scale for DSM-4 (CAPS-4) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-4. It contains symptom subscales, a CAPS-4 total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to Primary Endpoint (Primary Endpoint was approximately 18 weeks after Baseline and 1 month after the 2nd experimental session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 4
score on a scale | -21.5 (12.02) | -17.3 (13.05)

2. Secondary Outcome: Change in PTSD Diagnostic Scale (PDS) Total Severity Score From Baseline to Primary Endpoint
Description: The PTSD Diagnostic Scale (PDS) is a 49 item self-report measure designed to follow DSM-IV criteria for assessing PTSD. The PDS consists of a checklist to identify potentially traumatizing events experienced by the respondent and respondents then indicate which of the experienced events has troubled them the most in the last month and rate their response to this event at the time of its occurrence. Respondents then rate the severity of 17 items representing the cardinal symptoms of PTSD experienced in the past 30 days on a scale from 0 ("not at all") to 3 ("5 or more times a week") as well as the level of impairment caused by their symptoms across nine areas of life functioning. The 17 symptom severity items are summed to create a total symptom severity score, which ranges from 0 to 51, with higher scores indicating greater symptom severity and/or frequency.
Time Frame: as for outcome 1
Population: One participant in the MDMA group did not provide PDS data at Primary Endpoint so is excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 3
score on a scale | -1.0 (5.66) | -5.3 (1.53)

3. Secondary Outcome: Change in Beck Depression Inventory (BDI-II) Score From Baseline to Primary Endpoint
Description: The BDI-II is a validated 21-item self-report measure of symptoms of depression according to DSM-IV criteria. A BDI-II total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depressive symptoms. The scores range from 0 to 63, with higher score indicating greater severity of depressive symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 4
score on a scale | -4.0 (2.83) | 2.0 (15.34)

4. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Score From Baseline to Primary Endpoint
Description: The GAF Scale is a numeric scale ranging from 0 (serious risk of causing harm to the self or others) through 100 (superior function) that is used by mental health clinicians and physicians to subjectively rate the social, occupational, and psychological functioning of adults. The GAF is a reliable, validated measure of social functioning (Goldman, Skodol, and Lave, 1992). Higher scores indicate better functioning.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 4
score on a scale | 5.0 (4.24) | 5.3 (3.86)

5. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) Score From Baseline to Primary Endpoint
Description: The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances. It is comprised of 19 items that yield 7 component scores. Component scores are summed to create a total score. Total scores range from 0 (better) to 21 (worse), with higher scores indicating poor sleep quality.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 4
score on a scale | 1.0 (1.41) | -3.5 (3.32)

6. Secondary Outcome: Change in Dissociation Experiences Scale II (DES-II) Total Score From Baseline to Primary Endpoint
Description: The DES-II is a 28-item self-report measure of dissociation, defined as a lack of normal integration of an individual's thoughts, feelings, or experiences into the stream of consciousness or memory. It is an established measure of dissociative symptoms. The scale consists of statements describing facets of dissociation. Respondents indicate how often the specific experience happens to them, from from "never" (0% of the time) to "always" (100%). The scale is scored by treating percentages as single digits and averaging to produce a total score, ranging from 0 to 100. The higher the score, the more dissociative symptoms.
Time Frame: as for outcome 1
Population: DES-II data was not collected in one MDMA participant at the endpoint assessment so is excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 3
score on a scale | 8.4 (3.79) | -4.6 (13.63)

7. Secondary Outcome: Change in Posttraumatic Growth Inventory (PTGI) Total Score From Baseline to Primary Endpoint
Description: The PTGI is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains 5 subscales: relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life. Responses to each question are made on a scale of 0 (no change) to 5 (great degree of change), with higher scores indicating greater personal growth. Items are added to calculate the total PTGI score which ranges from 0 to 105, with higher scores indicative of greater growth.
Time Frame: as for outcome 1
Population: PTGI data was not collected in one MDMA participant at the endpoint assessment so is excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 3
score on a scale | 8.5 (14.85) | -3.7 (11.85)

ADVERSE EVENTS:
Time Frame: All AEs from baseline to the end of Stage 2 (approximately 10 months)
Description: Treatment group is the Stage 1 randomized treatment assignment (i.e. Results for "Placebo with Therapy" participants in Stage 2 reflect results following open-label crossover to complete 3 MDMA-assisted therapy sessions).
Groups:
- Placebo With Therapy (Stage 1): Participants will receive placebo during each of two experimental sessions.
  Placebo: Placebo administered in two experimental sessions; may take part in Stage 2 upon learning condition assignment
  Psychotherapy: Psychotherapy before and after experimental sessions
- MDMA-assisted Therapy (Stage 1): Participants will receive full-dose MDMA during each of two experimental sessions.
  3,4-methylenedioxymethamphetamine: Participants receive full-dose MDMA during two experimental sessions; after learning their condition assignment, participants will receive a third full-dose session.
  Psychotherapy: Psychotherapy before and after experimental sessions
- Placebo With Therapy (Stage 2): Stage 1 placebo participants will receive full-dose MDMA during each of two experimental sessions.
  3,4-methylenedioxymethamphetamine: Participants receive full-dose MDMA during two experimental sessions; after learning their condition assignment, participants will receive a third full-dose session.
  Psychotherapy: Psychotherapy before and after experimental sessions
- SRRs: Placebo With Therapy; SRRs: MDMA-assisted Therapy: Spontaneously reported reactions (SRRs) on blinded experimental session days and 7 days after.
Arm/Group | Placebo With Therapy (Stage 1) | MDMA-assisted Therapy (Stage 1) | Placebo With Therapy (Stage 2) | SRRs: Placebo With Therapy | SRRs: MDMA-assisted Therapy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 2/2 | 2/2 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Therapy (Stage 1) (N=2) | MDMA-assisted Therapy (Stage 1) (N=4) | Placebo With Therapy (Stage 2) (N=2) | SRRs: Placebo With Therapy (N=2) | SRRs: MDMA-assisted Therapy (N=4)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 4
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 2 | 4
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 2 | 4
Depressed Mood (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2 | 4
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Diarrhea (General disorders) | 0 | 0 | 0 | 0 | 2
Difficulty Concentrating (General disorders) | 0 | 0 | 0 | 2 | 3
Dizziness (General disorders) | 0 | 0 | 0 | 0 | 1
Dry mouth (General disorders) | 0 | 0 | 0 | 0 | 1
Impaired Gait/Balance (General disorders) | 0 | 0 | 0 | 0 | 2
Increased Irritability (General disorders) | 0 | 0 | 0 | 1 | 1
Jaw Clenching, Tight Jaw (General disorders) | 0 | 0 | 0 | 0 | 2
Lack of Appetite (General disorders) | 0 | 0 | 0 | 0 | 2
Low mood (General disorders) | 0 | 0 | 0 | 2 | 3
Muscle Tension (General disorders) | 0 | 0 | 0 | 2 | 3
Need More Sleep (General disorders) | 0 | 0 | 0 | 2 | 3
Perspiration (General disorders) | 0 | 0 | 0 | 1 | 2
Ruminations (General disorders) | 0 | 0 | 0 | 1 | 3
Sensitivity to Cold (General disorders) | 0 | 0 | 0 | 0 | 2
Weakness (General disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2014-06-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT01958593/Prot_003.pdf
  • Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT01958593/SAP_001.pdf
  • Informed Consent Form (2014-06-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT01958593/ICF_002.pdf